CLINICAL TRIAL: NCT05643794
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2A, Proof-Of-Concept Study to Evaluate the Efficacy and Safety of Rozanolixizumab to Treat Adult Study Participants With Severe Fibromyalgia Syndrome
Brief Title: A Proof-of-concept Study to Evaluate the Efficacy and Safety of Rozanolixizumab to Treat Adult Study Participants With Severe Fibromyalgia Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM0001
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
Keywords: Phase 2; Fibromyalgia; rozanolixizumab
MeSH Terms: conditions — Fibromyalgia | interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment sequence 1 (Experimental): Study participants on Treatment sequence 1 will receive rozanolixizumab and Placebo during the dosing period at pre-specified timepoints.
  Interventions: Drug: rozanolixizumab; Other: Placebo
- Treatment sequence 2 (Experimental): Study participants on Treatment sequence 2 will receive rozanolixizumab and Placebo during the dosing period at pre-specified timepoints.
  Interventions: Drug: rozanolixizumab; Other: Placebo
- Treatment sequence 3 (Placebo Comparator): Study participants on Treatment sequence 3 will receive Placebo during the dosing period at pre-specified timepoints.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: rozanolixizumab — Study participants will receive rozanolixizumab during the dosing periods as pre-defined.
  Other Names: UCB7665
  Arms: Treatment sequence 1; Treatment sequence 2
Other: Placebo — Study participants will receive Placebo during the dosing periods as pre-defined.
  Other Names: PBO

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of rozanolixizumab to treat adult study participants with severe fibromyalgia syndrome (FMS).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 years and ≤70 years of age at the time of signing the informed consent form (ICF)
* Study participant with a diagnosis of fibromyalgia as defined by the 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria (American College of Rheumatology Preliminary

Diagnostic Criteria) plus the following characteristics during the Screening Period:

1. Brief Pain Inventory-short form (BPI-SF) interference score ≥6.
2. Study participant has been diagnosed with fibromyalgia syndrome (FMS) for at least 6 months.
3. Study participant has been having FMS symptomatology for at least 2 years before enrollment - Capable of giving signed informed consent as described in the Protocol which includes compliance with the requirements and restrictions listed in the ICF and in the Study Protocol

Exclusion Criteria:

* Study participant has been diagnosed with fibromyalgia syndrome (FMS) for >15 years
* Study participant has any systemic autoimmune inflammatory disease
* Study participant has any medical or psychiatric or separate chronic pain condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study or the ability to assess FMS-related pain
* Study participant has severe renal impairment, defined as estimated glomerular filtration rate <30 mL/min/1.73 m^2, (calculated using Modification of Diet in Renal Disease [MDRD] study equation), at Screening visit
* Study participant has a clinically important active infection (including unresolved or not adequately treated infection) as assessed by the investigator
* Study participant has chronic inflammatory demyelinating polyneuropathy
* Study participant has a current or medical history of primary immunodeficiency
* Study participant is pregnant or lactating
* Study participant

  * Has suicide attempt in the past 2 years (including an active attempt, interrupted attempt, or aborted attempt),
  * OR had suicidal ideation with at least some intent to act in the past 6 months as indicated by a positive response (Yes) to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening or Baseline (Visit 3);
  * OR is otherwise judged clinically to be at a serious suicidal risk based on the investigator's judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (7):
- United Kingdom (7):
  - Fm0001 4405, Blackpool
  - Fm0001 4406, Cannock
  - Fm0001 4407, Leeds
  - Fm0001 4404, Liverpool
  - Fm0001 4402, Manchester
  - Fm0001 4403, Stockton-on-Tees
  - Fm0001 4401, Tankersley

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2022 and concluded in July 2024.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Sequence 1: RLZ 12w + RLZ 12w: Participants received placebo, subcutaneously (SC), once weekly (QW) for 2 weeks (Run-in Period), then rozanolixizumab (RLZ) 560 milligrams (mg), SC, QW, weekly (w) for 24 weeks (Treatment Period 1 + Treatment Period 2), followed by placebo SC, QW for 2 weeks (Runout Period). The safety follow-up (SFU) included all the participants who received the investigational medicinal product (IMP), regardless of discontinuation.
- Sequence 2: PBO + RLZ 12w: Participants received placebo SC, QW for 2 weeks (Run-in Period), then placebo SC, QW for 12 weeks (Treatment Period 1), followed by rozanolixizumab 560 mg, SC, QW for 12 weeks (Treatment Period 2), followed by placebo SC, QW for 2 weeks (Runout Period). The SFU included all the participants who received the IMP, regardless of discontinuation.
- Sequence 3: PBO + PBO: Participants received placebo SC, QW for 2 weeks (Run-in Period), then placebo SC, QW for 24 weeks (Treatment Period 1 + Treatment Period 2), followed by placebo SC, QW for 2 weeks (Run-out Period). The SFU included all the participants who received the IMP, regardless of discontinuation.
Period: Run-In (2 Weeks)
Arm/Group | Sequence 1: RLZ 12w + RLZ 12w | Sequence 2: PBO + RLZ 12w | Sequence 3: PBO + PBO
Started | 22 | 20 | 21
Completed | 22 | 20 | 21
Not Completed | 0 | 0 | 0
Period: Treatment Period 1 (12 Weeks)
Arm/Group | Sequence 1: RLZ 12w + RLZ 12w | Sequence 2: PBO + RLZ 12w | Sequence 3: PBO + PBO
Started | 22 | 20 | 21
Completed | 19 | 19 | 20
Not Completed | 3 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Consent Withdrawn by Study Participant (Not Due to Adverse Event) | 0 | 1 | 0
Period: Treatment Period 2 (12 Weeks)
Arm/Group | Sequence 1: RLZ 12w + RLZ 12w | Sequence 2: PBO + RLZ 12w | Sequence 3: PBO + PBO
Started | 19 | 19 | 20
Completed | 17 | 18 | 20
Not Completed | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Consent Withdrawn by Study Participant (Not Due to Adverse Event) | 1 | 0 | 0
Not completed — New Work Commitments | 1 | 0 | 0
Period: Run-Out Period (2 Weeks)
Arm/Group | Sequence 1: RLZ 12w + RLZ 12w | Sequence 2: PBO + RLZ 12w | Sequence 3: PBO + PBO
Started | 17 | 18 | 20
Completed | 17 | 18 | 20
Not Completed | 0 | 0 | 0
Period: Safety Follow-up Period (5 Weeks)
Arm/Group | Sequence 1: RLZ 12w + RLZ 12w | Sequence 2: PBO + RLZ 12w | Sequence 3: PBO + PBO
Started | 22 (The SFU included all the participants who received the IMP at any point in the study, regardless of treatment discontinuation.) | 20 (The SFU included all the participants who received the IMP at any point in the study, regardless of treatment discontinuation.) | 21 (The SFU included all the participants who received the IMP at any point in the study, regardless of treatment discontinuation.)
Completed | 22 | 20 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Set (RS) included all enrolled participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: RLZ 12w + RLZ 12w | Sequence 2: PBO + RLZ 12w | Sequence 3: PBO + PBO | Total
Number analyzed (Participants) | 22 | 20 | 21 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 20 | 61
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.9) | 47.8 (10.7) | 47.3 (9.5) | 47.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 17 | 55
  Male | 1 | 3 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 1 | 2
  White | 22 | 19 | 19 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 20 | 20 | 62

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Short Form (BPI-SF) Average Interference Score at 12 Weeks of Treatment
Description: The BPI-SF was a self-administered questionnaire used to evaluate the severity of a study participant's pain and the impact of this pain on the study participant's daily functioning. The BPI-SF assesses for the location of pain, pain intensity and functional interference from pain. The 7 BPI-SF interference items included: general activity, mood, walking ability, normal work (including housework), relations with other people, sleep, and enjoyment of life. Each item was rated on a 0 (did not interfere) to 10 (completely interfere) scale with a recall period of 24 hours. The BPI-SF interference score ranges 0-70. Higher scores indicated greater interference.
Time Frame: At 12 weeks of treatment
Population: Full Analysis Set (FAS) included all study participants who received any study treatment, including during the run-in period, had a baseline value and at least one post-baseline efficacy endpoint assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo (PBO): Participants received a PBO SC QW exposure up to 12 weeks and/or extended exposure from 12 to 24 weeks.
- RLZ 12 Weeks: Participants who received 12 weeks of RLZ 560 mg SC treatment during any sequence.
Arm/Group | Placebo (PBO) | RLZ 12 Weeks
Number analyzed (Participants) | 41 | 41
score on a scale | 6.30 [5.59 to 7.01] | 5.76 [5.11 to 6.41]
Statistical Analysis 1: Comparison: Placebo (PBO) vs RLZ 12 Weeks; Test type: Superiority; p = 0.129, Longitudinal linear mixed effect model; Difference from Placebo = -0.54, 95% CI 2-sided [-1.24 to 0.16] — The difference presented is RLZ 12 weeks minus Placebo

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE was defined as any AE with an onset date on or after the first dose of investigational medicinal product (IMP) in Run-In and on or before the earliest of the following: the last date of infusion (including Run-Out) +56 days, final contact date, or death. A TEAE is also defined as any unresolved event already present before administration of treatment that worsens in intensity following exposure to the treatment.
Time Frame: From Baseline till end of Safety Follow-up (up to Week 33)
Population: The Safety Set as treated (SS-t) included all study participants who received any study treatment, including during Run-In period.
Measure: Count of Participants; unit: Participants
Groups:
- Run-In-PBO: Participants received a PBO SC QW for 2 weeks in Run-In period. All study participants received placebo during the Run-in Period.
- TP1-RLZ: Participants received a RLZ 560 mg SC in Treatment Period 1 (TP1) up to Week 12.
- TP1-PBO: Participants received a PBO SC QW in TP1 up to Week 12. Pooled data is reported for placebo (Sequence 2 and Sequence 3).
- TP2-RLZ/RLZ: Participants who received RLZ in TP1 continued RLZ 560 mg SC in Treatment Period 2 (TP2) up to Week 24. One participant of "TP2-RLZ/RLZ" arm started TP2 but discontinued before receiving IMP.
- TP2-PBO/RLZ: Participants who received PBO in TP1 continued RLZ 560 mg SC in Treatment Period 2 (TP2) up to Week 24.
- TP2-PBO/PBO: Participants who received PBO in TP1 continued PBO SC in Treatment Period 2 (TP2) up to Week 24.
- Run-Out and SFU-RLZ/RLZ: Participants who received RLZ in TP1 and continued RLZ 560 mg SC up to Week 24 in TP2 received placebo SC, QW for 2 weeks in Run-Out period and had safety-follow-up (SFU), up to 5 weeks.
- Run-Out and SFU-PBO/RLZ: Participants who received PBO in TP1 and continued RLZ 560 mg SC up to Week 24 in TP2 received placebo SC, QW for 2 weeks in Run-Out period and had SFU, up to 5 weeks.
- Run-Out and SFU-PBO/PBO: Participants who received PBO in TP1 and continued PBO SC up to Week 24 in TP2 received placebo SC, QW for 2 weeks in Run-Out period and had SFU, up to 5 weeks.
Arm/Group | Run-In-PBO | TP1-RLZ | TP1-PBO | TP2-RLZ/RLZ | TP2-PBO/RLZ | TP2-PBO/PBO | Run-Out and SFU-RLZ/RLZ | Run-Out and SFU-PBO/RLZ | Run-Out and SFU-PBO/PBO
Number analyzed (Participants) | 63 | 22 | 41 | 18 | 19 | 20 | 22 | 20 | 21
Participants | 44 | 22 | 41 | 18 | 19 | 19 | 10 | 12 | 11

3. Secondary Outcome: Number of Participants With TEAEs Leading to Withdrawal of IMP
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE was defined as any AE with an onset date on or after the first dose of IMP in Run-In and on or before the earliest of the following: the last date of infusion (including Run-Out) +56 days, final contact date, or death.
Time Frame: From Baseline till end of Safety Follow-up (up to Week 33)
Population: The SS-t included all study participants who received any study treatment, including during Run-In period.
Measure: Count of Participants; unit: Participants
Groups:
- TP1-RLZ: Participants received RLZ 560 mg SC in TP1 up to Week 12.
- TP1-PBO: Participants received PBO SC QW in TP1 up to Week 12. Pooled data is reported for placebo (Sequence 2 and Sequence 3).
Arm/Group | Run-In-PBO | TP1-RLZ | TP1-PBO | TP2-RLZ/RLZ | TP2-PBO/RLZ | TP2-PBO/PBO | Run-Out and SFU-RLZ/RLZ | Run-Out and SFU-PBO/RLZ | Run-Out and SFU-PBO/PBO
Number analyzed (Participants) | 63 | 22 | 41 | 18 | 19 | 20 | 22 | 20 | 21
Participants | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 2

4. Secondary Outcome: Brief Pain Inventory Short Form (BPI-SF) Average Interference Score at 24 Weeks of Treatment
Description: as for outcome 1
Time Frame: At 24 weeks of treatment
Population: FAS included all study participants who received any study treatment, including during the run-in period, had a baseline value and at least one post-baseline efficacy endpoint assessment. Here 'overall number of participants analyzed' signifies participants evaluable for this Outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo: Participants received a PBO SC QW exposure up to 12 weeks and/or extended exposure from 12 to 24 weeks.
- RLZ 24 Weeks: Participants who received 24 weeks of RLZ 560 mg SC treatment during any sequence.
Arm/Group | Placebo | RLZ 24 Weeks
Number analyzed (Participants) | 41 | 18
score on a scale | 6.30 [5.59 to 7.01] | 5.79 [4.97 to 6.60]
Statistical Analysis 1: Comparison: Placebo vs RLZ 24 Weeks; Test type: Superiority; p = 0.358, Longitudinal mixed effects model; Difference from Placebo = -0.51, 95% CI 2-sided [-1.60 to 0.58] — The difference presented is RLZ 24 weeks minus PBO 24 weeks

5. Secondary Outcome: Revised Fibromyalgia Impact Questionnaire (FIQR) Score at 12 Weeks of Treatment
Description: The Revised Fibromyalgia Impact Questionnaire (FIQR) was a 21-item questionnaire with a recall period of 7 days. The FIQR included 3 domains: activities, overall impact, and symptoms. Each item was based on an 11-point numeric rating scale. The FIQR total score was calculated by taking the sum of the following: Activities domain subtotal divided by 3, overall impact" domain subtotal and symptoms domain subtotal divided by 2. The total score ranged from 0 to 100, with 0 denoting the best possible condition and 100 denoting the worst possible condition. Higher scores indicated more severe impact.
Time Frame: At 12 weeks of treatment
Population: FAS included all study participants who received any study treatment, including during the run-in period, had a baseline value and at least one post-baseline efficacy endpoint assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo (PBO) | RLZ 12 Weeks
Number analyzed (Participants) | 41 | 41
score on a scale | 70.70 [64.90 to 76.50] | 62.30 [57.32 to 67.28]
Statistical Analysis 1: Comparison: Placebo (PBO) vs RLZ 12 Weeks; Test type: Superiority; p = 0.003, Longitudinal mixed effects model; Difference from Placebo = -8.40, 95% CI 2-sided [-13.84 to -2.96] — The difference presented is RLZ 12 weeks minus Placebo

6. Secondary Outcome: Mean 7-day Average Daily Pain Score Assessed With Pain Numeric Rating Scale (NRS) at 12 Weeks of Treatment
Description: The Pain Numeric Rating Scale (NRS) was a scale in which a respondent selected a whole number that best described "How much pain have you experienced on average over the past 24 hours?" The 11-point Pain NRS ranged 0 (no pain) to 10 (pain as bad as you can imagine). Mean pain scores were derived the average of the daily assessment over the past 7 days. The higher score represented worst possible pain.
Time Frame: At 12 Weeks of treatment
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | RLZ 12 Weeks
Number analyzed (Participants) | 41 | 41
score on a scale | 6.59 [5.96 to 7.21] | 6.63 [6.09 to 7.18]
Statistical Analysis 1: Comparison: Placebo vs RLZ 12 Weeks; Test type: Superiority; p = 0.878, Longitudinal mixed effects model; Differences from Placebo = 0.05, 95% CI 2-sided [-0.55 to 0.64] — The differences presented is RLZ 12 weeks minus Placebo

7. Secondary Outcome: Mean 7-day Fatigue Score Assessed With Fatigue Numeric Rating Scale at 12 Weeks of Treatment
Description: The Fatigue Numeric Rating Scale (NRS) was a scale in which a respondent selected a whole number that best described "How much fatigue have you experienced on average over the past 24 hours?" The 11-point Fatigue NRS ranged 0 (no fatigue) to 10 (fatigue as bad as you can imagine). Mean fatigue scores were derived the average of the daily assessment over the past 7 days. Higher score represented worst possible fatigue.
Time Frame: At 12 weeks of treatment
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo (PBO) | RLZ 12 Weeks
Number analyzed (Participants) | 41 | 41
score on a scale | 7.26 [6.66 to 7.86] | 6.98 [6.45 to 7.51]
Statistical Analysis 1: Comparison: Placebo (PBO) vs RLZ 12 Weeks; Test type: Superiority; p = 0.352, Longitudinal mixed effects model; Difference from Placebo = -0.28, 95% CI 2-sided [-0.86 to 0.31] — The difference presented is RLZ 12 weeks minus Placebo

ADVERSE EVENTS:
Time Frame: From Baseline till end of Safety Follow-up (up to Week 33)
Description: TEAE: any AE with start date on or after first dose of IMP in Run-In, and on or before earliest of following: last date of infusion (including Run-Out, if applicable) +56 days, final contact date or death. TEAE also defined as any unresolved event already present before administration of treatment that worsens in intensity following exposure to treatment. The SS-t included all study participants who received any study treatment, including during Run-In period.
Arm/Group | Run-In-PBO | TP1-RLZ | TP1-PBO | TP2-RLZ/RLZ | TP2-PBO/RLZ | TP2-PBO/PBO | Run-Out and SFU-RLZ/RLZ | Run-Out and SFU-PBO/RLZ | Run-Out and SFU-PBO/PBO
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/22 | 0/41 | 0/18 | 0/19 | 0/20 | 0/22 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/22 | 3/41 | 0/18 | 0/19 | 0/20 | 0/22 | 1/20 | 2/21
Other Adverse Events (participants affected / at risk) | 24/63 | 21/22 | 37/41 | 18/18 | 19/19 | 16/20 | 3/22 | 8/20 | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In-PBO (N=63) | TP1-RLZ (N=22) | TP1-PBO (N=41) | TP2-RLZ/RLZ (N=18) | TP2-PBO/RLZ (N=19) | TP2-PBO/PBO (N=20) | Run-Out and SFU-RLZ/RLZ (N=22) | Run-Out and SFU-PBO/RLZ (N=20) | Run-Out and SFU-PBO/PBO (N=21)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In-PBO (N=63) | TP1-RLZ (N=22) | TP1-PBO (N=41) | TP2-RLZ/RLZ (N=18) | TP2-PBO/RLZ (N=19) | TP2-PBO/PBO (N=20) | Run-Out and SFU-RLZ/RLZ (N=22) | Run-Out and SFU-PBO/RLZ (N=20) | Run-Out and SFU-PBO/PBO (N=21)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (7) | 3 (4) | 1 (2) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (13) | 9 (14) | 17 (22) | 4 (5) | 7 (7) | 3 (4) | 0 (0) | 4 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (13) | 4 (9) | 4 (5) | 3 (5) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site urticaria (General disorders) | 0 (0) | 1 (12) | 0 (0) | 1 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 4 (4) | 0 (0) | 5 (13) | 0 (0) | 2 (6) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 4 (7) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type IV hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 6 (8) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 6 (8) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mammary duct ectasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT05643794/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT05643794/SAP_001.pdf